CLINICAL TRIAL: NCT06571591
Title: A Multicentre, Randomized, Double-blind, Placebo-controlled, Phase III Study to Evaluate the Efficacy and Safety of Pioglitazone Co-administration in Patients With Type II Diabetes With Insufficient Glycemic Control With Metformin and Empagliflozin Combination Therapy
Brief Title: Efficacy and Safety of Pioglitazone Combination Therapy in Type 2 Diabetes Patients on a Background of Empagliflozin With Metformin
Acronym: CT-L03
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT-L03-301; CT-L03 (Other: celltrion Inc.)
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: T2DM
MeSH Terms: interventions — empagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Active Comparator)
  Interventions: Drug: CT-L03 Group 1; Drug: Empagliflozin; Drug: Metformin
- Group 2 (Active Comparator)
  Interventions: Drug: CT-L03 Group 2; Drug: Empagliflozin; Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: Empagliflozin; Drug: Metformin

INTERVENTIONS:
Drug: CT-L03 Group 1 — tablets, QD, oral administration
  Arms: Group 1
Drug: CT-L03 Group 2 — tablets, QD, oral administration
  Arms: Group 2
Drug: Placebo — tablets, QD, oral administration
  Arms: Placebo
Drug: Empagliflozin — tablet, QD, oral administration
Drug: Metformin — tablets, oral administration

SUMMARY:
Phase 3 study to assess the Efficacy and Safety of CT-L03-301 in Type 2 Diabetes Patients with Insufficient Glycemic Control with Metformin and Empagliflozin Combination Therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults at the time of signing the Informed Consent Form (ICF)
* Signed the written ICF voluntarily after being fully informed of the objectives, methods, and effects of the study
* Diagnosed with T2DM

Exclusion Criteria:

* Diagnosed with other types of diabetes than T2DM
* History of hypersensitivity reaction to the components or drugs of the same class as the IP or the background therapy
* Uncontrolled severe complications of diabetes

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Week 24 of the Treatment
  Change from Baseline in HbA1c

SECONDARY OUTCOMES:
HbA1c | Week 12 of the Treatment
  Change from Baseline in HbA1c
FPG | Week 12 and 24 of the Treatment
  Change from Baseline in fasting plasma glucose
Body weight | Week 12 and 24 of the Treatment
  Change from Baseline in body weight

CONTACTS AND LOCATIONS:
Locations (1):
- Celltrion, Incheon, South Korea